CLINICAL TRIAL: NCT01373177
Title: A Randomized Crossover Study to Evaluate Differences Between the Bayley-II and the Bayley-III in Very Preterm Infants at 2 Years
Brief Title: Differences Between the Bayley-II and the Bayley-III in Very Preterm Infants at 2 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 10-007937
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Infant Development

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSID-II, then Bayley-III (Active Comparator): Receive BSID-II testing 4-8 weeks before Bayley-III testing
  Interventions: Diagnostic Test: Bayley Scales of Infant Development-II; Diagnostic Test: Bayley Scales of Infant Development-III
- Bayley-III, then BSID-II (Active Comparator): Receive Bayley-III testing 4-8 weeks before BSID-II testing
  Interventions: Diagnostic Test: Bayley Scales of Infant Development-II; Diagnostic Test: Bayley Scales of Infant Development-III

INTERVENTIONS:
Diagnostic Test: Bayley Scales of Infant Development-II — Individually administered test, designed to evaluate the developmental functioning of infants and small children, between 1 and 42 months of age. The purpose of the test is to identify infants and children with developmental delay. BSID-II was published in 1993. BSID-II provides normative data from two scales - Mental Development Index (MDI), and Psychomotor Development Index (PDI).
  Other Names: BSID-II
Diagnostic Test: Bayley Scales of Infant Development-III — Individually administered test, designed to evaluate the developmental functioning of infants and small children, between 1 and 42 months of age. The purpose of the test is to identify infants and children with developmental delay. BSID-III was released in 2006. BSID-III provides normative data from five scales - Cognitive, Language, Motor, Social-Emotional, and Adaptive.
  Other Names: Bayley-III; BSID-III

SUMMARY:
The objective of this randomized study is to test the hypothesis that scores on the Bayley Scales of Infant Development-III (Bayley-III) are higher than scores on the Bayley Scales of Infant Development-II (BSID-II) in the same group of infants who were born very preterm.

DETAILED DESCRIPTION:
The objective of this randomized crossover study is to test the hypothesis that scores on the Bayley Scales of Infant Development-III are higher than scores on the Bayley Scales of Infant Development-II in the same group of infants who were born very preterm. First, however, the investigators must demonstrate that significant "learning" does not occur when the tests are administered 4-8 weeks apart. The investigators hypothesize that scores on the Bayley-III will be higher than scores on the BSID-II, irrespective of the order in which the tests are administered.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <2000 grams and <32 weeks
* Corrected age of 18-22 months.

Exclusion Criteria:

* English is not the primary language in the child's home.
* Parent is unable to give informed consent for research participation.
* Parent is unable to commit to returning for follow-up testing in 4-8 weeks.
* Infant has severe medical illness or disability expected to impact his/her ability to participate in testing (ex: blindness, deafness, severe cerebral palsy, autism, tracheostomy).
* No exclusion for economic status, gender, race or ethnicity.
* Participation in a RCT that restricts timing and administration of developmental testing.

Ages: 18 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the mean difference between BSID-II Mental Development Index (MDI) and Bayley-III Cognitive Score. | 18-22 months

SECONDARY OUTCOMES:
Mean difference between BSID-II Physical Development Index and Bayley-III Composite Motor Score. | 18-22 months
Proportion of infants classified as having "developmental delay" (MDI <70 on BSID-II or either Language or Cognitive Score <70 on the Bayley-III). | 18-22 months
The mean difference in scores between time point one and time point two (a measure of learning or training). | 18-22 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara B. DeMauro, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States